CLINICAL TRIAL: NCT05541562
Title: A Practical Nomogram Based on Systemic Inflammatory Markers for Predicting Portal Vein Thrombosis in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYW2LL26362
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Systemic Inflammatory Markers; Portal Vein Thrombosis
Keywords: Portal Vein Thrombosis; systemic inflammatory markers
MeSH Terms: interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PVT group: The diagnosis of LC was based on clinical, laboratory, and radiological analyses, and/or liver biopsies. PVT was diagnosed according to the consensus for management of PVT in LC (2020, Shanghai) [1]. The inclusion criteria were as follows: (I) age ≥18 years, (II) Doppler ultrasound was the first-choice imaging modality; however, enhanced computed tomography or magnetic resonance imaging could also be used for confirmation at the time of admission to our hospital, and (III) patients with PVT on imaging examination but with insufficient evidence for the diagnosis of cirrhosis, hepatic vein pressure gradient measurement, and liver biopsy. Patients with primary or secondary hepatic malignant tumors, other malignant tumors, hematologic diseases, Budd-Chiari syndrome, non-cirrhotic PVT, inflammatory diseases, and other severe diseases were excluded.
  Interventions: Diagnostic Test: clinical laboratory tests, and imaging characteristics
- Non-PVT group: (1) Patients with cirrhosis diagnosed in accordance with the 2019 Guidelines for the Diagnosis and Treatment of Cirrhosis;(2)Color ultrasound, CT, MRI, and other imaging studies confirmed the absence of portal vein thrombosis and the specific location of the thrombosis.
  Interventions: Diagnostic Test: clinical laboratory tests, and imaging characteristics

INTERVENTIONS:
Diagnostic Test: clinical laboratory tests, and imaging characteristics — Data included the demographic status, etiology of the liver disease, clinical laboratory tests, and imaging characteristics. Clinical laboratory tests included D-dimer, activated partial thromboplastin time (APTT), prothrombin time (PT), antithrombin III, international normalized ratio (INR), thrombin time (TT), albumin (Alb), serum creatinine, hemoglobin, platelet count, white blood cell count, neutrophil count, lymphocyte count, monocyte count, model for end-stage liver disease (MELD) score, and Child-Pugh score. Imaging characteristics included splenic vein diameter, splenic vein velocity, portal vein diameter, and portal vein velocity.

SUMMARY:
Immunothrombosis has recently been used to describe the responses/mechanisms in thrombosis. Systemic inflammatory markers are prognostic markers for a variety of thrombotic conditions; however, their potential value in predicting portal vein thrombosis (PVT) is unknown. This study aimed to establish an easy-to-use nomogram based on systemic inflammatory markers to predict portal vein thrombosis (PVT) in patients with liver cirrhosis.

DETAILED DESCRIPTION:
This retrospective study included 478 patients with cirrhosis between January 2013 and January 2021. Reputed systemic inflammatory markers (systemic immune-inflammation index [SII], neutrophil-to-lymphocyte ratio [NLR], monocyte-to-lymphocyte ratio [MLR], and platelet-to-lymphocyte ratio (PLR)) were measured, and the clinical data were recorded. The independent risk factors for PVT were determined using univariate analyses and multivariate logistic regression analyses, and a nomogram to predict the occurrence of PVT was established. The concordance index, receiver operating characteristic curves, and calibration plots were used to evaluate the performance of the model.

ELIGIBILITY:
Inclusion Criteria:The diagnosis of LC was based on clinical, laboratory, and radiological analyses, and/or liver biopsies. PVT was diagnosed according to the consensus for management of PVT in LC (2020, Shanghai) [1]. The inclusion criteria were as follows: (I) age ≥18 years, (II) Doppler ultrasound was the first-choice imaging modality; however, enhanced computed tomography or magnetic resonance imaging could also be used for confirmation at the time of admission to our hospital, and (III) patients with PVT on imaging examination but with insufficient evidence for the diagnosis of cirrhosis, hepatic vein pressure gradient measurement, and liver biopsy. -

Exclusion Criteria:Patients with primary or secondary hepatic malignant tumors, other malignant tumors, hematologic diseases, Budd-Chiari syndrome, non-cirrhotic PVT, inflammatory diseases, and other severe diseases were excluded.

-

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study included 478 patients with cirrhosis between January 2013 and January 2021 at the Affiliated Hospital of Qingdao University (China).There were 239 patients with portal vein thrombosis and 239 patients without portal vein thrombosis.
Sampling Method: Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
systemic inflammatory markers | 9 years
  systemic immune-inflammation index [SII], neutrophil-to-lymphocyte ratio [NLR], monocyte-to-lymphocyte ratio [MLR], and platelet-to-lymphocyte ratio (PLR)

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No